CLINICAL TRIAL: NCT00059683
Title: Vaginal Ultrasound Cerclage Trial
Brief Title: Ultrasound-indicated Cerclage to Prevent Premature Birth in High-risk Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John Owen, Professor Ob/Gyn-Maternal Fetal medicine, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U01HD039939-01A1 (NIH)
Record Dates: First submitted 2003-05-01; First posted 2003-05-05 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Labor, Premature
Keywords: Preterm Birth; Premature Birth; Cervical cerclage; Vaginal ultrasound; Cervical length
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical Cerclage Group (Experimental): Women randomized to receive cerclage should receive cervical cerclage
  Interventions: Procedure: cervical cerclage
- Control Group (No Intervention): Women randomized to not receive cerclage represent the control arm

INTERVENTIONS:
Procedure: cervical cerclage — Cerclage is a circumferential stitch of non-absorbable suture placed around the cervix
  Arms: Cervical Cerclage Group

SUMMARY:
Pregnant women who have a shortened cervix and have previously had a premature baby are at increased risk for having another premature baby. This study will determine whether reinforcing the cervix with a surgical stitch can reduce the chance of a premature birth.

DETAILED DESCRIPTION:
Women with a prior early spontaneous preterm birth and a shortened mid-trimester cervical length (less than 25 mm) are at very high risk for having another premature baby. The Vaginal Ultrasound Cerclage Trial is a multicenter, randomized clinical trial designed to determine the efficacy of cerclage (a purse-string suture placed around the uterine cervix) for the prevention of spontaneous preterm birth prior to 35 weeks' gestation. The study will evaluate women at significant risk for recurrent spontaneous preterm birth (those with a prior spontaneous birth at 17 to 32 weeks' gestation) and who have an increased risk based on mid-trimester ultrasound findings of a cervical length less than 25 mm.

The trial will have an observational portion and an interventional portion. In the observational portion, 1,000 women with a history of a spontaneous preterm birth at 17 to 32 weeks' gestation will undergo biweekly vaginal ultrasounds beginning at 16 to 18 weeks' gestation and ending by 22 weeks. Prior research indicates that one third of these women will either have or develop a cervix less than 25 mm long. Women will be seen at a frequency determined by the cervical length (as determined by ultrasound examination starting at 16 weeks' gestation). If cervical length remains greater than 30 mm, the next visits will occur in 2 week intervals until 22.6 weeks' gestation. If the cervical length is 25 mm to 29 mm, the visits will be scheduled weekly. If the cervical length shortens to less than 25 mm, the woman is eligible for randomization, and will undergo one more study visit.

In the interventional portion of the trial, women will be randomized to either cerclage or no cerclage (control group). Randomized women will have weekly contact with a nurse either by phone or in person, whichever is convenient for the woman, until delivery occurs. The woman is followed during the course of her pregnancy and delivery of her infant. Her infant is followed until discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria

* Pregnant with a singleton gestation
* History of at least 1 prior spontaneous preterm birth at or before 32 weeks' gestation

Exclusion Criteria

* Cervical cerclage planned for this pregnancy
* Clinical history of cervical incompetence
* Untreated C. trachomatis or N. gonorrhoeae infection or symptomatic vaginitis
* Unable to obtain mid-trimester ultrasound to confirm no major fetal anomaly (i.e., aneuploidy, major organ system defect) or fetal demise prior to enrollment
* Multiple gestation
* Prolapsed or ruptured membranes noted on initial speculum examination
* Cervical os dilation > 2 cm noted on initial speculum examination
* Oligohydramnios
* Complete placenta previa
* Chronic hypertension or vascular disease requiring therapy
* Maternal red cell alloimmunization
* Insulin dependent diabetes
* Significant renal or cardiopulmonary disease
* Delivery or prenatal care outside clinical center
* Enrolled in this study in a previous pregnancy
* Participation in a randomized trial with interventions or endpoints in conflict with the cerclage randomized trial

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2003-01; Primary Completion 2007-11 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Incidence of preterm birth less than 35 weeks' gestation | Birth

SECONDARY OUTCOMES:
Gestational age at birth | birth

CONTACTS AND LOCATIONS:
Overall Officials: John Owen, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Owen J, Hankins G, Iams JD, Berghella V, Sheffield JS, Perez-Delboy A, Egerman RS, Wing DA, Tomlinson M, Silver R, Ramin SM, Guzman ER, Gordon M, How HY, Knudtson EJ, Szychowski JM, Cliver S, Hauth JC. Multicenter randomized trial of cerclage for preterm birth prevention in high-risk women with shortened midtrimester cervical length. Am J Obstet Gynecol. 2009 Oct;201(4):375.e1-8. doi: 10.1016/j.ajog.2009.08.015. PMID 19788970